CLINICAL TRIAL: NCT02095509
Title: Plasma Anti-FXa Concentration After Continuous Intravenous Infusion and Subcutaneous Dosing of Enoxaparin for Thromboprophylaxis in Critically Ill Patients
Brief Title: Pharmacokinetics of Enoxaparin in Intensive Care Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tampere University Hospital (Other)
Collaborators: Helsinki University Central Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2012-004599-21
Record Dates: First submitted 2014-03-18; First posted 2014-03-24 (Estimated); Last update posted 2017-10-27 (Actual); Status verified 2017-10

CONDITIONS: Venous Thromboembolism
MeSH Terms: conditions — Venous Thromboembolism | interventions — Enoxaparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Subcutaneous Enoxaparin (Active Comparator): Subcutaneous enoxaparin 40 mg every 24 hours for three days
  Interventions: Drug: Enoxaparin
- Intravenous Enoxaparin (Active Comparator): 40 mg enoxaparin daily as continuous intravenous infusion for three days (72 hours)
  Interventions: Drug: Enoxaparin

INTERVENTIONS:
Drug: Enoxaparin — Drug class: Low-molecular weight heparin
  Other Names: Klexane (sanofi-Aventis Oy, Finland)

SUMMARY:
To evaluate the pharmacokinetics of the thromboprophylactic agent enoxaparin in critically ill patients by comparing plasma anti-factor Xa activity when enoxaparin is administered either as a continuous intravenous infusion or subcutaneous bolus once daily.

To investigate possible ongoing coagulation by coagulation markers during antithrombotic therapy with standard doses of enoxaparin

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index between 18-30 kg/m2
* Critically ill patients requiring intensive care and pharmacological thromboprophylaxis
* Expected to remain in the ICU for at least 72 h
* Written informed consent obtained from the patient or his/her legal representative.

Exclusion Criteria:

* Other indications for anticoagulant therapy than thromboprophylaxis
* Intracranial haemorrhage or central neurosurgical operation within three months prior to the admission
* Disseminated intravascular coagulation (DIC) according to the international society on Thrombosis and Haemostasis criteria
* Known heparin induced thrombocytopenia (HIT), or hypersensitivity to enoxaparin or heparin
* Treatment with enoxaparin or any other low-molecular weight heparin (LMWH) or heparin within 24 hours prior to ICU admission. If patient has received thromboprophylactic dose of LMWH within 24-72 hours before ICU admission inclusion can be done if measured anti-factor Xa level is <0.1 IU/ml at the time of admission
* Any long-term anticoagulant medication, expect low-dose aspirin
* Major bleeding within the last week unless definitively treated
* Blood platelet count <50, P-thromboplastin time (TT) <40% , international normalized ratio (INR) >1.7
* Glomerular filtration rate less than 50 ml/min/1.73 m2 estimated from serum creatinine by applying Cockcroft-Gault equation or chronic dialysis
* HIV, hepatitis B virus, or hepatitis C virus infection
* Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2014-03; Primary Completion 2016-06-30 (Actual); Study Completion 2016-09-30 (Actual)

PRIMARY OUTCOMES:
Plasma anti-factor Xa level | 72 hours
  Change in plasma anti-factor Xa levels between baseline and 72 hours

SECONDARY OUTCOMES:
Incidence of Venous thromboembolism | 90 days
  If clinically suspected a compression ultrasound will be done
Incidence of Bleeding | 90 days
  Major and minor bleeding events will be reported

CONTACTS AND LOCATIONS:
Locations (2):
- Finland (2):
  - Tampere University Hospital, Tampere, Pirkanmaa
  - Helsinki University Central Hospital, Meilahti, Helsinki, Uusimaa